CLINICAL TRIAL: NCT01619332
Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of LEZ763 Following Single and Multiple Ascending Doses in Healthy Subjects and Patients With Type 2 Diabetes
Brief Title: Clinical Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of LEZ763
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLEZ763X2201
Record Dates: First submitted 2012-06-12; First posted 2012-06-14 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2016-03

CONDITIONS: Type II Diabetes
Keywords: Healthy volunteers,; Diabetes; Glucose; Pharmacokinetics
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- LEZ763 (Experimental): Part I- Healthy volunteers enrolled into 6 single-ascending dose cohorts Part II- Healthy volunteers enrolled into 5 multiple-ascending dose cohorts. Part III- LEZ763 will be given orally once daily for 28 days in a randomized and blinded manner
  Interventions: Drug: LEZ763
- Placebo (Placebo Comparator): Part I : Healthy volunteers enrolled in 6 single ascending dose cohorts to receive matching placebo of LEZ763. Part II: Healthy volunteers enrolled in 5 multiple ascending dose cohorts to receive matching placebo of LEZ763. Part III- Placebo will be given orally once daily for 28 days to patients assigned to placebo in a randomized and blinded manner
  Interventions: Drug: Placebo
- Sitagliptin (Active Comparator): Sitaglitpin will be given orally once daily for 28 days to patients assigned to this treatment in a randomized and blinded manner
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: Placebo — Placebo will be given orally once daily for 28 days to patients assigned to placebo in a randomized and blinded manner
  Arms: Placebo
Drug: Sitagliptin — Sitaglitpin will be given orally once daily for 28 days to patients assigned to this treatment in a randomized and blinded manner
  Arms: Sitagliptin
Drug: LEZ763 — LEZ763 will be given orally once daily for 28 days in a randomized and blinded manner
  Arms: LEZ763

SUMMARY:
This study is a three part study to assess the safety and efficacy of LEZ763 on normal healthy volunteers and patients with Type 2 Diabetes.

ELIGIBILITY:
Inclusion criteria:

* All subjects: (suggest this will reduce duplication)
* Male or female aged 18-65 yr,
* Subjects must weigh at least 50 kg to participate in the study. Body mass index (BMI) must be within the range of 18-37 kg/m2 (inclusive
* Only postmenopausal females or female subjects who report surgical sterilization (women without child bearing potential) will be allowed in this study.
* Subjects with stable conventional sleep-wake cycle

Normal Healthy Volunteers

* Healthy male or female subjects,
* must be in good health (as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at Screening).

Type II Diabetic Patients

* Type 2 diabetes diagnosed by American Diabetes Association criteria for at least 3 months prior to screening.
* Patients either drug naïve or on stable dose of metformin (stable dose for at least 4 weeks prior to Screening). The metformin dose should remain constant during the course of the study.
* HbA1c 6.5 to 9.5 % inclusive at screening

Exclusion criteria:

All subjects:

* Smokers (use of tobacco products in the previous 3 months).
* Donation or loss of 400 mL or more of blood within 8 weeks prior to first dosing, or longer if required by local regulation.
* Significant illness within two weeks prior to dosing.
* Have (or have history of) drug or alcohol abuse within the 12 months prior to dosing or evidence of such abuse as indicated by the laboratory assays conducted during the screening or baseline evaluations

Normal Healthy Volunteers

• History of diabetes, or adrenal disorders.

Type II Diabetic Patients

* Type 1 diabetes mellitus; positive anti-GAD antibodies; acquired or secondary forms of diabetes such as those resulting from pancreatic surgery/injury, cystic fibrosis related diabetes
* Evidence of clinically significant diabetic complications (such nephropathy, retinopathy, neuropathy) Other protocol defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2012-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Number of Patients with adverse events, serious adverse events and death | Day 28
  An adverse event is the appearance or worsening of any undesirable sign, symptom, or medical condition occurring after starting the study drug even if the event is not considered to be related to study drug. Adverse events will also be determined on the basis of clinical laboratory assessments, electrocardiographic evaluations and vital signs determinations.
Pharmacokinetics of LEZ763 (Part I): area under the plasma concentration-time curve from time zero to infinity (AUCinf) | pre-dose, and 0.5, 0.66, 0.75, 1, 1.5, 2, 2.5, 3, 3.5 4, 6, 8, 12 hours post-dose on Day 1; 24 and 36 hours Day 2; Day 3, Day 4
  Blood will be collected at multiple timepoints and will be analyzed for LEZ736 concentrations after single dose
Pharmacokinetics of LEZ763 (Part I): area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration (AUClast) | pre-dose, and 0.5, 0.66, 0.75, 1, 1.5, 2, 2.5, 3, 3.5 4, 6, 8, 12 hours post-dose on Day 1; 24 and 36 hours Day 2; Day 3, Day 4
  Blood will be collected at multiple timepoints and will be analyzed for LEZ736 concentrations after single dose
Pharmacokinetics of LEZ763 (Part I): Terminal elimination half-life (T1/2) | pre-dose, and 0.5, 0.66, 0.75, 1, 1.5, 2, 2.5, 3, 3.5 4, 6, 8, 12 hours post-dose on Day 1; 24 and 36 hours Day 2; Day 3, Day 4
  Blood will be collected at multiple timepoints and will be analyzed for LEZ736 concentrations after single dose
Pharmacokinetics of LEZ763 (Part I): Apparent systemic (or total body) clearance from plasma following extravascular administration (CL/F) | pre-dose, and 0.5, 0.66, 0.75, 1, 1.5, 2, 2.5, 3, 3.5 4, 6, 8, 12 hours post-dose on Day 1; 24 and 36 hours Day 2; Day 3, Day 4
  Blood will be collected at multiple timepoints and will be analyzed for LEZ736 concentrations after single dose
Pharmacokinetics of LEZ763 (Part I) : Observed maximum plasma concentration (Cmax) following drug administration | pre-dose, and 0.5, 0.66, 0.75, 1, 1.5, 2, 2.5, 3, 3.5 4, 6, 8, 12 hours post-dose on Day 1; 24 and 36 hours Day 2; Day 3, Day 4
  Blood will be collected at multiple timepoints and will be analyzed for LEZ736 concentrations after single and multiple doses
Pharmacokinetics of LEZ763 (Part I): time to reach the maximum concentration after drug administration (Tmax) | pre-dose, and 0.5, 0.66, 0.75, 1, 1.5, 2, 2.5, 3, 3.5 4, 6, 8, 12 hours post-dose on Day 1; 24 and 36 hours Day 2; Day 3, Day 4
  Blood will be collected at multiple timepoints and will be analyzed for LEZ736 concentrations after single dose
Pharmacokinetics of LEZ763 (Part II) : Observed maximum plasma concentration (Cmax) following drug administration | pre-dose, and 0.5, 0.66, 0.75, 1, 1.5, 2, 2.5, 3, 3.5 4, 6, 8, 12 hours post-dose on Day 1 and Day 10
  Blood will be collected at multiple timepoints and will be analyzed for LEZ736 concentrations after multiple doses
Pharmacokinetics of LEZ763 (Part II): time to reach the maximum concentration after drug administration (Tmax) | pre-dose, and 0.5, 0.66, 0.75, 1, 1.5, 2, 2.5, 3, 3.5 4, 6, 8, 12 hours post-dose on Day 1 and Day 10
  Blood will be collected at multiple timepoints and will be analyzed for LEZ736 concentrations after multiple doses
Pharmacokinetics of LEZ763 (Part II): Accumulation ratio(Racc) | pre-dose, and 0.5, 0.66, 0.75, 1, 1.5, 2, 2.5, 3, 3.5 4, 6, 8, 12 hours post-dose on Day 1 and Day 27
  Blood will be collected at multiple timepoints and will be analyzed for LEZ736 concentrations after multiple doses
Pharmacokinetics of LEZ763 (Part III) : Observed maximum plasma concentration (Cmax) following drug administration | pre-dose, and 0.5, 0.66, 0.75, 1, 1.5, 2, 2.5, 3, 3.5 4, 6, 8, 12 hours post-dose on Day 1 and Day 27
  Blood will be collected at multiple timepoints and will be analyzed for LEZ736 concentrations after multiple doses
Pharmacokinetics of LEZ763 (Part III): time to reach the maximum concentration after drug administration (Tmax) | pre-dose, and 0.5, 0.66, 0.75, 1, 1.5, 2, 2.5, 3, 3.5 4, 6, 8, 12 hours post-dose on Day 1 and Day 27
  Blood will be collected at multiple timepoints and will be analyzed for LEZ736 concentrations after multiple doses
Pharmacokinetics of LEZ763 (Part III): Area under the plasma concentration-time curve from time zero to the end of the dosing interval tau (AUCtau) | pre-dose, and 0.5, 0.66, 0.75, 1, 1.5, 2, 2.5, 3, 3.5 4, 6, 8, 12 hours post-dose on Day 1 and Day 27
  Blood will be collected at multiple timepoints and will be analyzed for LEZ736 concentrations after single and multiple doses
Pharmacokinetics of LEZ763 (Part III): Accumulation ratio(Racc) | pre-dose, and 0.5, 0.66, 0.75, 1, 1.5, 2, 2.5, 3, 3.5 4, 6, 8, 12 hours post-dose on Day 1 and Day 27
  Blood will be collected at multiple timepoints and will be analyzed for LEZ736 concentrations after single and multiple doses
Pharmacokinetics of LEZ763 and Sitagliptin (Part III): Observed maximum plasma concentration (Cmax) following drug administration | pre-dose, and 0.5, 0.66, 0.75, 1, 1.5, 2, 2.5, 3, 3.5 and 4 hours post-dose on Day 28
  Blood will be collected at multiple timepoints and will be analyzed for LEZ736 concentrations after multiple doses
Pharmacokinetics of LEZ763 and Sitagliptin (Part III): Area under the plasma concentration-time curve from time zero to the end of the dosing interval tau (AUCtau) | pre-dose, and 0.5, 0.66, 0.75, 1, 1.5, 2, 2.5, 3, 3.5 and 4 hours post-dose on Day 28
  Blood will be collected at multiple timepoints and will be analyzed for LEZ736 concentrations after multiple doses
Pharmacokinetics of LEZ763 and Sitagliptin (Part III): Time to reach the maximum concentration after drug administration (Tmax) | pre-dose, and 0.5, 0.66, 0.75, 1, 1.5, 2, 2.5, 3, 3.5 and 4 hours post-dose on Day 28
  Blood will be collected at multiple timepoints and will be analyzed for LEZ736 concentrations after multiple doses
Area under the effect curve (AUC0-4h) over the 4-hour post-dose period to measure glucose response following a standard mixed meal test | 4 hour post-dose Day 27

SECONDARY OUTCOMES:
Area under the serum Glucagon-like-peptide 1 (GLP-1) curve (AUC0-24 hours) | Pre-dose, and 0.5, 0.66, 0.75, 1, 1.5, 2, 2.5, 3, 3.5 and 4 hours post-dose on Day -1, Day 1, Day 27, and Day 28
  GLP-1 Biomarker measures will be evaluated at pre-dose, and 0.5, 0.66, 0.75, 1, 1.5, 2, 2.5, 3, 3.5 and 4 hours post-dose
2-hour value of post-prandial glucose | Day 1 of Part I, Day 1 and day 10 of Part II
Change from baseline in Fasting C-peptide at Day 27 (Part III) | Baseline, Day 27
Change from baseline in Fasting Insulin at Day 27 (Part III) | Baseline , Day 27
Change from baseline in fasting plasma glucose at Day 27 (Part III) | Baseline , Day 27
Change From Baseline in peak glucose level following meal Test at Day 27 (Part III) | Baseline , Day 27
Peak effect (Emax) on postprandial GLP-1 (Part III) | Baseline , Day 27
Change from baseline in Peptide YY (PYY) (Part III) | Baseline , Day 27
Change from baseine in Gastric inhibit polypeptide (GIP) (Part III) | Baseline , Day 27

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- United States (6):
  - Novartis Investigative Site, Chula Vista, California
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Knoxville, Tennessee
  - Novartis Investigative Site, San Antonio, Texas

REFERENCES:
- See also: Results for CLEZ763X2201 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=12503